CLINICAL TRIAL: NCT02509130
Title: MISSION Severe Asthma: Modern Innovative Solutions to Improve Outcomes in Severe Asthma. A Mixed Methods Observational Comparison of Clinical Outcomes in MISSION Versus Current Care Delivery.
Brief Title: MISSION Severe Asthma Modern Innovative Solutions to Improve Outcomes in Severe Asthma.
Acronym: MISSION
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2015/15
Record Dates: First submitted 2015-07-13; First posted 2015-07-27 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
Keywords: Severe Asthma; Asthma; Specialised Asthma Care; Asthma Care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patients who attended RAAC/SAAC.: Patients who have previously attended the Rapid Access Asthma Clinic (RAAC) will be approached for the quantitative study. Patients who went onto the attend the Severe Asthma Assessment Clinics (SAAC) will also be approached for the quantitative and qualitive parts of the study.
- Patients eligible for RAAC, but DNA'd: Patients identified by the GP search, who did not attend the previous MISSION clinics will be approached to participate in the quantitative part of the study.
- Asthma Outpatients: Patients who are attending outpatient clinics as new referrals will be approached to participate in the quantitative part of the study.
- Healthcare Professionals: Healthcare professionals who performed the MISSION RAAC or SAAC will be approached for qualitative interview part of the study only.

SUMMARY:
MISSION is a new and novel way of delivering highly specialised asthma care and has the potential to change the way asthma care across the United Kingdom (UK) is delivered as well as services for other long term health conditions. The MISSION model is the first model of this type and the current research study aims to evaluate its success and to compare the MISSION service to current care delivery. This will be done in several different ways. The study is a mixed methods evaluation of the new service comparing outcomes before and after the intervention using retrospective data analysis and prospective qualitative interview. A control arm of patients not exposed to, but eligible for, the new intervention will also be included. The study will be conducted at Portsmouth Hospitals National Health Service (NHS) Trust and will recruit patients who attended MISSION clinics, outpatient asthma clinics, staff who attended MISSION clinics in a professional capacity and patients from GP surgeries where MISSION clinics were held who did not attend.

DETAILED DESCRIPTION:
Purpose and design

The purpose of the study is to evaluate in detail the clinical and health economic outcomes from the MISSION project. The MISSION clinics combined a new way of delivering asthma care along with actively case finding patients who were not already known to specialist services but who had uncontrolled or at risk asthma.

The aim of the study is to compare the MISSION clinic model outcomes to current clinic model outcomes as well as performing qualitative interviews with patients who attended and staff who took part in the project.The research study was developed by a team from Portsmouth Hospital Trust and the University of Portsmouth including a research fellow, consultant and Professor, research methodologist, qualitative senior lecturer and independent statistician. A patient adviser also reviewed the lay summary and patient information sheets. The study undergoes independent review by another clinician as part of the sponsor process.

The study is also part of an MD project for the University of Portsmouth.

Design:

This is a mixed methods study.

A quantitative analysis of data from patients who attended the MISSION Rapid Access Asthma Clinics (RAAC), patients who attended the MISSION Severe Asthma Assessment Clinics (SAAC), patients who were invited to the RAAC but did not attend and patients who have been referred by their GP to the severe asthma clinic during the same time MISSION was running. The data analysis will include asthma control, hospital admissions, GP appointments, related medical conditions,medications, investigations and assessments done and time between appointments.

A qualitative study will be conducted using telephone interviews with patients who attended the SAAC and health care professionals who took part in the MISSION clinics.

The aim is to recruit:

* 44 MISSION patients (of whom 20 attended both the RAAC and the SAAC),
* 132 patients who were invited to MISSION RAAC but did not attend
* 20 patients referred to the severe asthma clinic at the hospital
* 20 health care professionals who took part in the MISSION clinics

Methodology:

Participants will be approached for consent by post. They will be given time to read the information and return the consent form to the study team. They will be given a contact number to discuss any questions.

Once a participant has consented to the quantitative study there is no further study procedures for the participant. Participants will be asked for consent to collect data from their GP and hospital records for the study. This will be entered onto a form (CRF) against a study number and then into a password protected study database held on a secure server at Portsmouth Hospitals NHS Trust. This data will then be analysed by a statistician and research fellow.

Participants for qualitative interview will have an interview over the telephone lasting 45 minutes to one hour. This will be recorded and transcribed. The participant will be given the transcript to read and correct. The transcripts will then be analysed looking for themes.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Is in one of the following population groups:
* Attended the MISSION RAAC or
* Attended the MISSION SAAC or
* Identified as uncontrolled asthma by record searches and invited to MISSION RAAC but did not attend - 'primary care patients' or
* Has been referred to the specialist asthma clinic at Queen Alexandra Hospital - 'outpatient severe asthma patients' or
* Attended the MISSION RAAC or SAAC as a health care professional
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* The patient is unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with uncontrolled or potentially severe asthma identified from GP records by the MISSION team and new referrals to an asthma specialist clinic at Queen Alexandra Hospital between May and August 2014.
  Study participants for qualitative interview will be recruited from patients who attended MISSION SAAC days and staff who attended MISSION RAAC or SAAC days.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Asthma control as measured by exacerbation frequency for all patients | 6 months
  The primary endpoint is asthma control as measured by exacerbation frequency (defined as deterioration in symptoms requiring ≥30mg prednisolone or equivalent for ≥3 days) for all patients

SECONDARY OUTCOMES:
Short acting bronchodilator (SABA) use | 6 months
  Short acting bronchodilator (SABA) use measured by number of inhalers prescribed in 6 months pre and post MISSION SAAC, RAAC or outpatient clinic.
Exacerbation frequency | 6 months
  Exacerbation frequency (defined as deterioration in symptoms requiring ≥30mg prednisolone or equivalent for ≥3 days) in 6 months pre and post MISSION SAAC, RAAC or outpatient clinic.
Health care usage costs for asthma and number of contacts | 6 months
  Health care usage costs for asthma and number of contacts (GP visits, Emergency Department (ED) or out of hour attendances (OOH), hospital admissions, emergency GP visits) over 6 months pre and post MISSION or outpatient clinic.
Assessment of co-morbidity | 6 months
  Assessment of comorbidity (rhinosinusitis, anxiety and depression, dysfunctional breathing, gastro oesophageal reflux and obstructive sleep apnoea) and method of assessment for MISSION SAAC patients and outpatient severe asthma clinic patients
Assessment of inhaler technique and recommendations for inhaler devices. | 6 months
  Assessment of inhaler technique and recommendations for inhaler devices for MISSION SAAC patients and outpatient severe asthma clinic patients
Smoking cessation advice. | 6 months
  Smoking cessation advice for MISSION SAAC patients and outpatient severe asthma clinic patients
Investigations performed in secondary care | 6 months
  Investigations performed during 6 months in secondary care e.g. full lung function, sputum induction, High-Resolution Computed Tomography (HRCT) chest for MISSION SAAC patients and outpatient severe asthma clinic patients
Time from GP referral to 1st clinic visit | 6 months
  Time from GP referral to 1st clinic visit in secondary care for MISSION SAAC patients and outpatient severe asthma clinic patients
Time between 1st and 2nd visit | 6 months
  Time between 1st and 2nd visit in secondary care for MISSION SAAC patients and outpatient severe asthma clinic patients
Time to appointment with other specialists | 6 months
  Time to appoint with other specialists for asthma related comorbidity where indicated, e.g. dietician, Ear, Nose & Throat (ENT), physiotherapists, psychologist, CT imaging for MISSION SAAC patients and outpatient severe asthma clinic patients
Fractional Exhaled Nitric Oxide (FeNO) Assessment | 6 months
  Assessment of eosinophilic airways inflammation by FeNO for MISSION SAAC patients and outpatient severe asthma clinic patients
Frequency of non-attendance | 6 months
  The frequency of non-attendance at clinic for MISSION SAAC patients and outpatient severe asthma clinic patients
Severity of co-morbidities | 6 months
  Severity of co-morbidities for MISSION RAAC patients
Frequency of co-morbidities | 6 months
  Frequency of co-morbidities for MISSION RAAC patients
Frequency & type of allergy | 6 months
  Frequency & type of allergy for MISSION RAAC patients
Measurement of exhaled nitric oxide | 6 months
  Measurement of exhaled nitric oxide for MISSION RAAC patients
Measurement & variation of lung function (Single | 6 months
  Composite measurement & variation of lung function for MISSION RAAC patients
Frequency and type of additional asthma control medication. | 6 months
  Frequency and type of additional asthma control medication for MISSION RAAC patients
Quality of life | 6 months
  Quality of life as assessed by the Asthma Quality of Life Questionnaire (AQLQ).
Disease control | 6 months
  Disease control as assessed by the Asthma Control Questionnaire (ACQ)
Number of Forced Expiratory Volume at one second (FEV1) / Forced Vital Capacity (FVC) measurements | 6 months
  Number of patients having measurements of FEV1/FVC as a proxy for asthma control and severity in the MISSION RAAC patient and primary care patients
Prescription of SABA's | 6 months previous
  Prescription of Short Acting Bronchodilators (SABAs) during last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Prescription of SABA's | Baseline
  Prescription of Short Acting Bronchodilators (SABAs) during last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Prescription of SABA's | 6 months
  Prescription of Short Acting Bronchodilators (SABAs) during last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Exacerbation rates | 6 months previous
  Exacerbation rates (defined as deterioration in symptoms requiring ≥30mg prednisolone or equivalent for ≥3 days) during the last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Exacerbation rates | Baseline
  Exacerbation rates (defined as deterioration in symptoms requiring ≥30mg prednisolone or equivalent for ≥3 days) during the last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Exacerbation rates | 6 months
  Exacerbation rates (defined as deterioration in symptoms requiring ≥30mg prednisolone or equivalent for ≥3 days) during the last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
ED attendances during the last 6 months | 6 months previous
  Emergency Department (ED) attendances during the last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Out Of Hours (OOH) contacts during the last 6 months | 6 months previous
  Out Of Hours (OOH) contacts during the last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
Hospital admissions during the last 6 months | 6 months previous
  Emergency Department (ED) attendances, Out Of Hours (OOH) contacts and hospital admissions during the last 6 months at baseline and 6 months for MISSION RAAC and primary care patients.
ED attendances at baseline | Baseline
  Emergency Department (ED) attendances at baseline for MISSION RAAC and primary care patients.
OOH contacts at baseline | Baseline
  Out Of Hours (OOH) contacts at baseline for MISSION RAAC and primary care patients.
Hospital admissions at baseline | Baseline
  Hospital admissions at baseline for MISSION RAAC and primary care patients.
ED attendances at 6 months. | 6 months
  Emergency Department (ED) attendances at 6 months for MISSION RAAC and primary care patients.
Out Of Hours (OOH) contacts at 6 months | 6 months
  Out Of Hours (OOH) contacts at 6 months for MISSION RAAC and primary care patients.
Hospital admissions during at 6 months | 6 months
  Hospital admissions during at 6 months for MISSION RAAC and primary care patients.
Inhaled steroid doses and usage | 6 months
  Inhaled steroid doses and usage for MISSION RAAC and primary care patients.
sensitivity and specificity of the Primary Care Information Services (PRIMIS) Asthma Audit Tool | 6 months
  The sensitivity and specificity of the PRIMIS Asthma Audit Tool in identifying the patients compared to gold standard specialist assessment and interrogation of primary care records for MISSION RAAC and primary care patients.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Anoop J Chauhan, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

REFERENCES:
- [Background] Hoddinott P, Pill R. Qualitative research interviewing by general practitioners. A personal view of the opportunities and pitfalls. Fam Pract. 1997 Aug;14(4):307-12. doi: 10.1093/fampra/14.4.307. PMID 9283852
- [Background] Hoddinott P, Pill R. A review of recently published qualitative research in general practice. More methodological questions than answers? Fam Pract. 1997 Aug;14(4):313-9. doi: 10.1093/fampra/14.4.313. PMID 9283853
- [Background] Bulpitt H, Martin PJ. Who am I and what am I doing? Becoming a qualitative research interviewer. Nurse Res. 2010;17(3):7-16. doi: 10.7748/nr2010.04.17.3.7.c7741. PMID 20450084
- [Background] Richards H, Emslie C. The 'doctor' or the 'girl from the University'? Considering the influence of professional roles on qualitative interviewing. Fam Pract. 2000 Feb;17(1):71-5. doi: 10.1093/fampra/17.1.71. PMID 10673494
- See also: Asthma UK — http://www.asthma.org.uk
- See also: Department of Health - An outcomes strategy for people with chronic obstructive pulmonary disease (COPD) and asthma in England — http://www.gov.uk/government/publications/an-outcomes-strategy-for-people-with-chronic-obstructive-pulmonary-disease-copd-and-asthma-in-england
- See also: Five year forward view, NHS England — http://www.england.nhs.uk/wp-content/uploads/2014/10/5yfv-web.pdf